CLINICAL TRIAL: NCT01681225
Title: EPVent 2- A Phase II Study of Mechanical Ventilation Directed by Transpulmonary Pressures (EPVent2)
Brief Title: EPVent 2- A Phase II Study of Mechanical Ventilation Directed by Transpulmonary Pressures
Acronym: EPVent2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Daniel Talmor, Edward Lowenstein Professor of Anaesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009P000374; UM1HL108724 (NIH)
Record Dates: First submitted 2012-09-05; First posted 2012-09-07 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS; mechanical ventilation; ALI; esophageal pressure
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EPVent (Experimental): The overall goals for the "EPVent" group (esophageal-pressure guided mechanical ventilation) are to employ an open-lung strategy that includes low tidal volumes and maintenance of a positive transpulmonary pressure at end-expiration [Ptpexp]. Fraction of inspired oxygen [FiO2] and transpulmonary pressure pressure during an expiratory hold will be changed to achieve values shown in one of the columns of a protocol-specified table to meet the oxygenation target.
  Interventions: Other: Esophageal-pressure guided mechanical ventilation
- Control (Active Comparator): The overall goals for the Control group are similar to those for the EPVent group: to employ an open-lung strategy that includes low tidal volumes using an alternative high positive end-expiratory pressure [PEEP] strategy. The control group PEEP and tidal volume will be managed without reference to the esophageal pressure measurements, and instead will follow an empiric high PEEP mechanical ventilation strategy. PEEP and FiO2 will be raised or lowered to achieve the oxygenation target level specified in a study table.
  Interventions: Other: High PEEP mechanical ventilation

INTERVENTIONS:
Other: Esophageal-pressure guided mechanical ventilation
  Other Names: mechanical ventilation strategy; open-lung strategy; EPVent; positive transpulmonary pressure at end-expiration
  Arms: EPVent
Other: High PEEP mechanical ventilation
  Arms: Control

SUMMARY:
This phase II multi-centered, randomized controlled trial of mechanical ventilation directed by esophageal pressure measurement will test the primary hypothesis that using a strategy of maintaining a minimal but positive transpulmonary pressure (Ptp = airway pressure minus pleural pressure) throughout the ventilatory cycle will lead to an improvement in patient survival.

DETAILED DESCRIPTION:
This phase II prospective randomized controlled trial of ventilation directed by esophageal pressure measurements will enroll 200 patients with moderate to severe ARDS by the Berlin conference definition in several academic medical centers in North America. The control group will be ventilated using an alternative high-PEEP strategy with PEEP and FiO2 set using to an empiric table.

Plasma samples will be obtained at enrollment and days 3 and 7 and assessed for a variety of lung injury biomarkers to better assess the association between our intervention and the inflammation associated with mechanical ventilation and the development of ARDS. Hospital survivors will undergo a brief follow up phone survey to assess survival, functional status (Barthel Index), health-related QOL (Short Form 12), and frailty (VES) twelve months after enrollment.

The study length will be six years with a six month start-up period followed by a planned 50 month enrollment and twelve month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Acute onset of ARDS as defined by the Berlin Consensus Conference definitions:

  1. Hypoxemic respiratory failure with PaO2 / FIO2 ratio < 200 mmHg
  2. b) Bilateral alveolar/interstitial infiltrates on chest x-ray, with opacities not present for more than 7 days
  3. Respiratory failure not fully explained by cardiac failure or fluid overload
  4. Intubation on controlled ventilation and receiving PEEP ≥ 5 cm H2O
* Age 16 years or older
* Duration of ARDS 36 hours or less from meeting final Berlin criterion.

Exclusion Criteria:

* Received mechanical ventilation more than 96 hours
* Recently treated or bleeding varices, esophageal stricture, hematemesis, esophageal trauma, recent esophageal surgery or other contraindication for nasogastric tube placement
* Severe coagulopathy (platelet count < 5000/microliter or INR > 4)
* History of lung transplantation
* Elevated intracranial pressure or conditions where hypercapnia-induced elevations in intracranial pressure should be avoided
* Evidence of active air leak from the lung
* not committed to full support
* Participation in other intervention trials for ARDS or for sepsis within the past 30 days.
* Neuromuscular disease that impairs ability to ventilate spontaneously
* Severe chronic liver disease, defined as Child-Pugh Score of ≥12
* Treating clinician refusal, or unwillingness to commit to controlled ventilation for at least 24 hours
* Inability to get informed consent from the patient or surrogate.
* Use of rescue therapies for prior to enrollment (e.g. nitric oxide, ECMO, prone positioning, high frequency oscillation). This does not exclude cases where these therapies were used as the initial mode of ventilation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2012-10-31 (Actual); Primary Completion 2017-10-12 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
A composite outcome of mortality and time off the ventilator at 28-days. | Day 28
  The trial will utilize a primary composite endpoint that incorporates death and days off the ventilator at 28 days in such a manner that death constitutes a more serious outcome. Every subject is compared to every other subject in the trial and assigned one number resulting from each comparison. Since mortality outcome is clinically more important, mortality takes precedence over days off the ventilator. The sum of scores for patients in the treatment group is compared to the sum of scores of subjects in the control group to form a test statistic by the Mann-Whitney technique.

SECONDARY OUTCOMES:
Ventilator free days to day 28 | Day 28
  Number of calendar days breathing unassisted.
mortality | Day 60
  Hospital and ICU mortality to day 60
lengths of stay | Day 60
  Hospital and ICU lengths of stay to days 28 and 60
biomarkers of lung injury | Day 7
  Plasma biomarkers of lung injury on enrollment and days 3 and 7 after enrollment
Survival | 1 year
  Mortality to 1 year
Need for rescue therapy | Day 28
  Rescue measures will be chosen according to the practice at the clinical site, and may include repeated recruitment maneuvers, prone positioning, nitric oxide, epoprostenol sodium, airway pressure release ventilation, high frequency ventilation, or ECMO.
Activities of daily living | 1 year
  Will assess via questionnaire (Barthel Index) done by phone at 1 year. Barthel Index scores range from 0-100, with 100 representing greatest independence of activities of daily living.
Self-reported health assessment | 1 year
  Will assess via questionnaire (12-Item Short-Form Health Survey [SF-12]) done by phone at 1 year. The SF-12 scores range from 0-100 points, with higher scores representing the highest level of health.
Frailty in patients age 65 and older | 1 year
  Will assess via questionnaire (Vulnerable Elders-13 Survey) done by phone at 1 year. VES scores range from 0-10 points, with higher scores representing greater risk.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Talmor, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (14):
- United States (10):
  - University of California at San Diego, La Jolla, California
  - Stanford University Medical Center, Stanford, California
  - Orlando Health, Orlando, Florida
  - Shock-Trauma University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Massachusets Medical Center, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Montefiore Medical Center, The Bronx, New York
- Canada (4):
  - Vancouver General Hospital, Vancouver, British Columbia
  - St Joseph's Healthcare, Hamilton, Ontario
  - University Health Network, Toronto, Ontario
  - Laval University, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rubenfeld GD, Caldwell E, Peabody E, Weaver J, Martin DP, Neff M, Stern EJ, Hudson LD. Incidence and outcomes of acute lung injury. N Engl J Med. 2005 Oct 20;353(16):1685-93. doi: 10.1056/NEJMoa050333. PMID 16236739
- [Background] Herridge MS, Cheung AM, Tansey CM, Matte-Martyn A, Diaz-Granados N, Al-Saidi F, Cooper AB, Guest CB, Mazer CD, Mehta S, Stewart TE, Barr A, Cook D, Slutsky AS; Canadian Critical Care Trials Group. One-year outcomes in survivors of the acute respiratory distress syndrome. N Engl J Med. 2003 Feb 20;348(8):683-93. doi: 10.1056/NEJMoa022450. PMID 12594312
- [Background] Briel M, Meade M, Mercat A, Brower RG, Talmor D, Walter SD, Slutsky AS, Pullenayegum E, Zhou Q, Cook D, Brochard L, Richard JC, Lamontagne F, Bhatnagar N, Stewart TE, Guyatt G. Higher vs lower positive end-expiratory pressure in patients with acute lung injury and acute respiratory distress syndrome: systematic review and meta-analysis. JAMA. 2010 Mar 3;303(9):865-73. doi: 10.1001/jama.2010.218. PMID 20197533
- [Background] Brower RG, Lanken PN, MacIntyre N, Matthay MA, Morris A, Ancukiewicz M, Schoenfeld D, Thompson BT; National Heart, Lung, and Blood Institute ARDS Clinical Trials Network. Higher versus lower positive end-expiratory pressures in patients with the acute respiratory distress syndrome. N Engl J Med. 2004 Jul 22;351(4):327-36. doi: 10.1056/NEJMoa032193. PMID 15269312
- [Background] Meade MO, Cook DJ, Guyatt GH, Slutsky AS, Arabi YM, Cooper DJ, Davies AR, Hand LE, Zhou Q, Thabane L, Austin P, Lapinsky S, Baxter A, Russell J, Skrobik Y, Ronco JJ, Stewart TE; Lung Open Ventilation Study Investigators. Ventilation strategy using low tidal volumes, recruitment maneuvers, and high positive end-expiratory pressure for acute lung injury and acute respiratory distress syndrome: a randomized controlled trial. JAMA. 2008 Feb 13;299(6):637-45. doi: 10.1001/jama.299.6.637. PMID 18270352
- [Background] Gattinoni L, Caironi P, Carlesso E. How to ventilate patients with acute lung injury and acute respiratory distress syndrome. Curr Opin Crit Care. 2005 Feb;11(1):69-76. doi: 10.1097/00075198-200502000-00011. PMID 15659948
- [Background] Talmor D, Sarge T, Malhotra A, O'Donnell CR, Ritz R, Lisbon A, Novack V, Loring SH. Mechanical ventilation guided by esophageal pressure in acute lung injury. N Engl J Med. 2008 Nov 13;359(20):2095-104. doi: 10.1056/NEJMoa0708638. Epub 2008 Nov 11. PMID 19001507
- [Background] Talmor D, Sarge T, O'Donnell CR, Ritz R, Malhotra A, Lisbon A, Loring SH. Esophageal and transpulmonary pressures in acute respiratory failure. Crit Care Med. 2006 May;34(5):1389-94. doi: 10.1097/01.CCM.0000215515.49001.A2. PMID 16540960
- [Background] Sarge T, Talmor D. Targeting transpulmonary pressure to prevent ventilator induced lung injury. Minerva Anestesiol. 2009 May;75(5):293-9. PMID 19412147
- [Background] Fish E, Novack V, Banner-Goodspeed VM, Sarge T, Loring S, Talmor D. The Esophageal Pressure-Guided Ventilation 2 (EPVent2) trial protocol: a multicentre, randomised clinical trial of mechanical ventilation guided by transpulmonary pressure. BMJ Open. 2014 Oct 6;4(9):e006356. doi: 10.1136/bmjopen-2014-006356. PMID 25287106
- [Result] Beitler JR, Sarge T, Banner-Goodspeed VM, Gong MN, Cook D, Novack V, Loring SH, Talmor D; EPVent-2 Study Group. Effect of Titrating Positive End-Expiratory Pressure (PEEP) With an Esophageal Pressure-Guided Strategy vs an Empirical High PEEP-Fio2 Strategy on Death and Days Free From Mechanical Ventilation Among Patients With Acute Respiratory Distress Syndrome: A Randomized Clinical Trial. JAMA. 2019 Mar 5;321(9):846-857. doi: 10.1001/jama.2019.0555. PMID 30776290
- [Derived] Santarisi A, Suleiman A, Redaelli S, von Wedel D, Beitler JR, Talmor D, Goodspeed V, Jung B, Schaefer MS, Baedorf Kassis E. Transpulmonary Pressure as a Predictor of Successful Lung Recruitment: Reanalysis of a Multicenter International Randomized Clinical Trial. Respir Care. 2025 Jan;70(1):1-9. doi: 10.1089/respcare.11736. PMID 39964867